CLINICAL TRIAL: NCT05160038
Title: Embodied Virtual Reality for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Bigna Lenggenhager, Principal Investigator, University of Zurich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmbVRpain
Record Dates: First submitted 2021-11-01; First posted 2021-12-16 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Complex Regional Pain Syndromes; Complex Regional Pain Syndrome Type I of the Upper Limb; Complex Regional Pain Syndrome I (CRPS I); Complex Regional Pain Syndrome I of Upper Limb; Complex Regional Pain Syndrome Type II; Complex Regional Pain Syndrome II of Upper Limb; Peripheral Nerve Injury Upper Limb; Osteoarthritis Hand; Osteoarthritis Finger
Keywords: virtual reality; embodiment; embodied pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy; Causalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bodily illusions (Experimental): Participants in the experimental group see a bodily illusion applied to their embodied virtual avatar.
  Interventions: Device: Embodied virtual reality
- No bodily illusions (No Intervention): Participants in the control group embody a virtual avatar, but without bodily illusions

INTERVENTIONS:
Device: Embodied virtual reality — An immersive headmounted display visually depicts a relaxing woods scene, coupled with a virtual avatar that either shows bodily illusions or no bodily illusions
  Arms: Bodily illusions

SUMMARY:
Virtual reality creates interactive, multimodal sensory stimuli that have demonstrated considerable success in reducing pain. Much research so far has focused on VR's ability to shift patients' attention away from pain; however, these methods provide only transient relief through means of distraction and therefore do not offer long-term analgesic remediation. An alternative and promising approach is to utilize VR as an embodied simulation technique, where virtual body illusions are employed as tools to improve body perception and produce potentially more enduring analgesia.

Disturbances in body perception (i.e., alterations in the way the body is perceived) are increasingly acknowledged as a pertinent feature of chronic pain, and include aberrations in perceived shape, size, or color that differ from objective assessment. The degree of body perception distortion positively correlates with pain, and prior interventions have evinced that treatments aimed at reducing body perception distortions correspondingly ameliorate pain. Several recent experimental research studies have demonstrated the analgesic efficacy of body illusions in a range of pain conditions.

Immersive VR multisensory feedback training signifies a promising new avenue for the potential treatment of chronic pain by supporting the design of targeted virtual environments to alter (distorted) body perceptions. Various illusions have been described to alter pain perception; however, they. Have not been directly compared to each other. The multimodal stimulus control of VR enables physical-to-virtual body transfer illusions, resulting in the feeling that the virtual body is one's own. These virtual body illusions can modulate body perception with ease and could therefore be used to alter the perceived properties of pain, consequently utilizing a virtual avatar to specifically shape interactive processing between central and peripheral mechanisms.

DETAILED DESCRIPTION:
With roughly 1 in 5 affected individuals, chronic pain is incredibly widespread on a global scale. Unfortunately, standard opioidergic treatment does not consistently provide adequate relief and is often tied to adverse events. As a novel and innovative approach in pain management, virtual reality (VR) creates interactive, multimodal sensory stimuli that have demonstrated considerable success in reducing pain. Much research has focused on VR's ability to shift patients' attention away from pain; however, these methods provide only transient relief through means of distraction and therefore do not offer long- term analgesic remediation. A different and promising therapeutic approach is to utilize VR as an embodied simulation technique, where virtual body illusions can be used to improve body perception and produce potentially more enduring analgesia.

Disturbances in body perception (i.e., alterations in the way the body is perceived) are increasingly acknowledged as a pertinent feature of chronic pain. Compared to healthy individuals, patients afflicted with chronic pain exhibit alterations in neural areas involved in body perception. Subjectively, patients with chronic pain report aberrations in body perception that include alterations in perceived shape, size, or color that differ from objective assessment (e.g., experiencing painful body parts as enlarged, twisted, or otherwise distorted. Furthermore, the degree of body perception distortion positively correlates with pain, where those in more severe pain also report more extensive body perception disturbances. Interestingly, interventions aimed at reducing body perception distortion correspondingly ameliorate pain, and several studies have evinced that modulating body perception with the use of (non-virtual) body illusions (i.e., multisensory modulations of perceived embodiment) can elicit significant and even sustained analgesia in patients with chronic pain. Distorted perceptions of the body therefore constitute a promising target for pain modulation. Recent experimental and clinical research has demonstrated the analgesic efficacy of body illusions in a range of chronic pain conditions, including (but not limited to) osteoarthritis (OA), complex regional pain syndrome (CRPS), and neuropathic pain. For example, illusory stretching of the hands in patients with OA reduced pain by 40%. Furthermore, pain relief following a single illusion has been shown to persist between several minutes up 10 weeks, suggesting that multiple sessions of body illusions could reduce cortical misrepresentation over time and lead to long-term analgesia.

Immersive VR multisensory feedback training signifies a promising new avenue for potential future approaches aimed at the management of chronic pain by supporting the design of targeted virtual environments to alter (distorted) body perceptions. The multimodal stimulus control of VR enables physical-to-virtual body transfer illusions, resulting in the feeling that the virtual body is one's own. These virtual body illusions can modulate body perception with ease and could therefore be used to alter the perceived properties of pain: disturbed body perception in patients with chronic pain can thereby be improved by adapting the virtual body in ways that would not be possible with the physical body. The current study can be classified as risk category A, since it entails only minimal risks and burdens (i.e., potential but unlikely transient dizziness and nausea in VR).

The investigators hypothesize that virtual reality will reduce pain intensity ratings from pre- to post-virtual reality session. However, it is expected that virtual body illusions will lead to stronger analgesia, since the virtual body illusions additionally aim to target and normalize body perception disturbances that are associated with chronic pain. While analgesia is expected immediately following the VR distraction in the control group, cumulative improvements or sustained analgesia, nor any improvements in body perception disturbances are not expected. Additionally, the investigators therefore also hypothesize that virtual body illusions, but not virtual distraction, will reduce body perception disturbances.

This single center project will consist of confirmatory quantitative research conducted on a national level. The use of virtual reality (i.e., virtual reality as a distraction versus embodiment modality) will be examined as a modulatory interventional tool for pain management in different pain conditions, including complex regional pain syndrome, peripheral nerve injury, and osteoarthritis. To this end, the control condition will consist of the thus far regularly employed virtual distraction (i.e., a relaxing virtual scene of a wooded area to distract participants from pain), in which they will be immersed over several sessions, versus an experimental condition, wherein participants will be able to both choose from several virtual body illusions to identify which one best reduces their pain and body perception disturbances, and be immersed in the preferred/chosen virtual body illusion of choice over several sessions.

Participants of each pain syndromes will be assigned to the experimental or control group in a sequential counterbalanced manner. Participants will be grouped together according to their pain condition, and then assigned to the experimental or control group in a sequential counterbalanced manner to assure that individuals from each pain condition are equally represented in both groups. No blinding procedures will be necessary, since the control and experimental groups are clearly discerned.

A virtual avatar of each gender will be configured to match the gender of the participants. A visuomotor tracking system will be used to track the movements of participants' arms, which will match the movements of the virtual body to increase illusory ownership of the virtual avatar. The Oculus Quest 2 (www.oculus.com) will be used to as an HMD for the virtual environments, which has 6GB of RAM and 1832 x 1920 pixels per eye. It weighs 503 grams, has a screen refresh rate of 72 Hz at launch, and uses internal cameras to track the limbs. The software for both the experimental and control group will be programmed in Unity (Unity Technologies, San Francisco); a commonly employed software for programming virtual scenarios (for empirical research).

Participants will be informed that the aim of the study is to compare the efficacy of virtual distraction versus virtual embodiment on pain perception, and that while both virtual distraction and virtual embodiment have demonstrated analgesic efficacy in the past, they will only be allocated to one of the groups. During the intervention, participants will be seated in a chair with both arms resting on a table in front of them and will first be familiarized with the virtual environment. In the virtual scene, they will experience a matching virtual table which will be located in a relaxing virtual scene matching the virtual scene of the control condition - i.e., a virtual scene of a forest, as well as a virtual body seen from a first-person perspective. Participants will be asked to move their arms from side to side to induce synchronous visuomotor tracking between the virtual and physical body and therefore induce illusory ownership of the virtual body.

During the first session of virtual body illusions, participants (both experimental and control groups) will first experiment with the different types of body illusions provided - i.e., stretching, shrinking, synchronous flashing of the virtual body with the heart rate, transparency, or blue color modification. The stretching illusion will consist of a normal arm or hand stretching beyond its physical boundaries, and then shrinking back to its normal state. In the shrinking illusion, the limb will shrink in size before increasing to a normal size again. Another illusion will include visual depiction of the heart rate, where the virtual body part will flash in synchrony with the heartbeat of the participant. The transparency condition will consist of a limb increasing and decreasing in transparency, while the color modification will include a limb that can be cooled through changing the color to blue. This will allow for an individualized approach, wherein participants in the experimental group can first experiment with and then move forward with the virtual illusion they perceive to most effectively reduce their pain. Participants in the control group will also complete these initial virtual body illusions to increase the statistical power to examine the effectiveness of the different types of virtual body illusions. To minimize carry-over effects, the different types of virtual body illusions will be presented in a counterbalanced manner. Each illusion will be presented for 45 seconds, which falls in line with previous research using body illusions for chronic pain.

Prior to each illusion, a pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). Each virtual body illusion will be presented three times, and after each illusion, another pain-intensity NRS will appear asking participants to rate their pain. Additionally, following each type of body illusion, participants will be asked to rate the degree of embodiment of the virtual avatar and their own body (embodiment questionnaire - long version: 1. How strongly did the participant feel that they were present in the virtual environment? 2. How much did the participant feel like the virtual arm is their own arm? 3. How strongly does it feel like the movements of the virtual arm are the participant's own movements? 4. How much does the participant feel like the virtual arm is a different person? 5. How much a part of their body does the participant's affected physical body part feel? 6. How aware is the participant of the physical position of their physical limb? 7. How much attention is the participant currently paying to their physical limb? 8. How strong are the emotional feelings that they have about their limb? Questions 5-8 are adapted from the Bath CRPS Body Perception Disturbance Scale. All questions will be answered on a visual analog scale (VAS) from 'not at all' to 'very much', except for question 8, which will be answered from 'very negative' to 'very positive'). Participants will be given a two-minute break between each different type of virtual body illusion.

After participants have chosen the virtual body illusion that most strongly reduces their pain intensity NRS, or the one they feel most comfortable with, they will be given a 15 minute break. Following the break, participants will begin the first session with their chosen virtual body illusion. The virtual body illusions will be presented in blocks, with one block consisting of 3 x 45 second virtual body illusion sessions. Between the 45 second virtual body illusions of each block, there will be a 10 second break from the body illusion. Prior to the first and following each block, participants will rate their pain on the pain intensity NRS. In total, participants will complete five blocks of virtual body illusions, with a 2 minute break between each block. After completion of all five blocks, participants will again complete the embodiment questionnaire, after which the HMD will be removed. In total, participants will spend about 20 minutes in virtual reality during the five blocks.

Participants in the control group will similarly be familiarized with the HMD and virtual reality, and will also complete the baseline in which they will experience the same virtual body illusions as the experimental group, and report their pain intensity NRS. Following the VR intro session, they will also be given a 15 minute break. Participants in the control group will not continue with virtual body illusions; instead, they will only be exposed to the relaxing virtual scene with no body shown, which will be identical between the control and experimental group. Participants will answer the pain-intensity NRS at comparable time intervals to the experimental group, therefore similarly completing one pre pain-intensity NRS prior to beginning the virtual reality distraction session, and 5 "post" pain-intensity NRS. Therefore, participants in the control condition will spend a similar amount of time (approximately 20 minutes) in virtual reality. Similarly, they will also complete an embodiment questionnaire, except a shorter version that will not include questions 2-4 of the embodiment questionnaire - longer version, and instead will only assess the body perceptions of their physical bodies (embodiment questionnaire - short version: 1. How strongly did the participant feel that they were present in the virtual environment? 2. How much a part of their body does their affected physical body part feel? 3. How aware is the participant of the physical position of their physical limb? 4. How much attention is the participant currently paying to their physical limb? 5. How strong are the emotional feelings that they have about their limb?).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by the participants
* Presence of one of the following chronic pain conditions of the upper limbs:

osteoarthritis (OA), complex regional pain syndrome (CRPS)

Exclusion Criteria:

* Inability to follow study procedures, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
* Extreme motion sickness, nausea, or dizziness to the virtual simulations
* Currently pregnant or breastfeeding women
* High risk populations for Covid-19 (i.e., high blood pressure, chronic respiratory condition, diabetes, presence of autoimmune disease, cardiovascular disease, presence of cancer)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Pain assessment baseline | through study completion, an average of 2 weeks
  A first pain assessment will be made at baseline. A pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). The pain intensity NRS during the VR sessions will be answered within the virtual environment, where questions will be presented to participants within the headmounted display (HMD), which participants can then answer using a cursor that is controlled by head movements.
Pain assessment post - block 1 (session 1 - 4) | through study completion, an average of 2 weeks
  Pain assessment will be made after the first block of VR, which lasts about 140 seconds. A pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). The pain intensity NRS during the VR sessions will be answered within the virtual environment, where questions will be presented to participants within the headmounted display (HMD), which participants can then answer using a cursor that is controlled by head movements.
Pain assessment post - block 2 (session 1 - 4) | through study completion, an average of 2 weeks
  Pain assessment will be made after the second block of VR, which lasts about 140 seconds. A pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). The pain intensity NRS during the VR sessions will be answered within the virtual environment, where questions will be presented to participants within the headmounted display (HMD), which participants can then answer using a cursor that is controlled by head movements.
Pain assessment post - block 3 (session 1 - 4) | through study completion, an average of 2 weeks
  Pain assessment will be made after the third block of VR, which lasts about 140 seconds. A pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). The pain intensity NRS during the VR sessions will be answered within the virtual environment, where questions will be presented to participants within the headmounted display (HMD), which participants can then answer using a cursor that is controlled by head movements.
Pain assessment post - block 4 (session 1 - 4) | through study completion, an average of 2 weeks
  Pain assessment will be made after the fourth block of VR, which lasts about 140 seconds. A pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). The pain intensity NRS during the VR sessions will be answered within the virtual environment, where questions will be presented to participants within the headmounted display (HMD), which participants can then answer using a cursor that is controlled by head movements.
Pain assessment post - block 5 (session 1 - 4) | through study completion, an average of 2 weeks
  Pain assessment will be made after the fifth block of VR, which lasts about 140 seconds. A pain-intensity numeric rating scale (NRS) will appear with the written instruction asking participants to judge the intensity of their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). The pain intensity NRS during the VR sessions will be answered within the virtual environment, where questions will be presented to participants within the headmounted display (HMD), which participants can then answer using a cursor that is controlled by head movements.

SECONDARY OUTCOMES:
Body perception disturbances - post VR session 1 | through study completion, an average of 2 weeks
  Participants provide answers to their current body perception (experimental and control groups), as well as to the embodiment of the avatar (experimental group only). The embodiment questionnaire during the VR session will be administered within the virtual environment in the HMD, which participants can then answer using a cursor that is controlled by head movements.
Body perception disturbances - post VR session 2 | through study completion, an average of 2 weeks
  Participants provide answers to their current body perception (experimental and control groups), as well as to the embodiment of the avatar (experimental group only). The embodiment questionnaire during the VR session will be administered within the virtual environment in the HMD, which participants can then answer using a cursor that is controlled by head movements.
Body perception disturbances - post VR session 3 | through study completion, an average of 2 weeks
  Participants provide answers to their current body perception (experimental and control groups), as well as to the embodiment of the avatar (experimental group only). The embodiment questionnaire during the VR session will be administered within the virtual environment in the HMD, which participants can then answer using a cursor that is controlled by head movements.
Body perception disturbances - post VR session 4 | through study completion, an average of 2 weeks
  Participants provide answers to their current body perception (experimental and control groups), as well as to the embodiment of the avatar (experimental group only). The embodiment questionnaire during the VR session will be administered within the virtual environment in the HMD, which participants can then answer using a cursor that is controlled by head movements.
Pain ratings for each bodily illusion during session 1 - bodily illusion 1 | through study completion, an average of 2 weeks
  All participants (experimental and control group) will complete a first session in which they try out the five different bodily illusions (counterbalanced order). The first pain rating will be collected following the first bodily illusion.
Pain ratings for each bodily illusion during session 1- bodily illusion 2 | through study completion, an average of 2 weeks
  All participants (experimental and control group) will complete a first session in which they try out the five different bodily illusions (counterbalanced order). The second pain rating will be collected following the second bodily illusion.
Pain ratings for each bodily illusion during session 1- bodily illusion 3 | through study completion, an average of 2 weeks
  All participants (experimental and control group) will complete a first session in which they try out the five different bodily illusions (counterbalanced order). The third pain rating will be collected following the third bodily illusion.
Pain ratings for each bodily illusion during session 1- bodily illusion 4 | through study completion, an average of 2 weeks
  All participants (experimental and control group) will complete a first session in which they try out the five different bodily illusions (counterbalanced order). The fourth pain rating will be collected following the fourth bodily illusion.
Pain ratings for each bodily illusion during session 1- bodily illusion 5 | through study completion, an average of 2 weeks
  All participants (experimental and control group) will complete a first session in which they try out the five different bodily illusions (counterbalanced order). The fifth pain rating will be collected following the fifth bodily illusion.

OTHER OUTCOMES:
VR side effects - session 1 | through study completion, an average of 2 weeks
  After each VR session, participants will be asked whether they experienced any negative side effects, such as dizziness or nausea, and will be asked to rate and describe their experiences in VR - both positive and negative. Participants will also be asked to rate their mood and relaxation they experienced during the VR sessions.
VR side effects - session 2 | through study completion, an average of 2 weeks
  After each VR session, participants will be asked whether they experienced any negative side effects, such as dizziness or nausea, and will be asked to rate and describe their experiences in VR - both positive and negative. Participants will also be asked to rate their mood and relaxation they experienced during the VR sessions.
VR side effects - session 3 | through study completion, an average of 2 weeks
  After each VR session, participants will be asked whether they experienced any negative side effects, such as dizziness or nausea, and will be asked to rate and describe their experiences in VR - both positive and negative. Participants will also be asked to rate their mood and relaxation they experienced during the VR sessions.
VR side effects - session 4 | through study completion, an average of 2 weeks
  After each VR session, participants will be asked whether they experienced any negative side effects, such as dizziness or nausea, and will be asked to rate and describe their experiences in VR - both positive and negative. Participants will also be asked to rate their mood and relaxation they experienced during the VR sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland